CLINICAL TRIAL: NCT02303418
Title: Carbetocin Versus Oxytocin in the Prevention of Post Partum Haemorrhage (PPH) in Women Undergoing Caesarean Sections for Placenta Previa: A Randomised Controlled Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PPH1
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Post Partum Haemorrhage
Keywords: Obstetrics
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbetocin (Active Comparator): 100 µgm of Carbetocin will be diluted in 10ml saline and will be given by the anesthesist slowly intravenously after delivery of the baby. The uterine tone and amount of bleeding will be noted and the need for further uterotonic agents will be determined 2 minutes after giving the drug.
  Interventions: Drug: Carbetocin
- Oxytocin (Active Comparator): 5 mg of oxytocin will be diluted in 10ml saline and will be given by the anesthesist slowly intravenously after delivery of the baby. The uterine tone and amount of bleeding will be noted and the need for further uterotonic agents will be determined 2 minutes after giving the drug.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Carbetocin — Carbetocin will be given slowly iv after delivery of the baby
  Arms: Carbetocin
Drug: Oxytocin — Oxytocin will be given slowly iv after delivery of the baby
  Arms: Oxytocin

SUMMARY:
The study aims at comparing the roles of carbetocin and oxytocin in the prevention of atonic PPH in women undergoing CS for placenta previa.

200 women will be randomly divided into 2 equal groups using computer generated random numbers, Group 1 will receive Carbetocin 100 µgm (Pabal® Ferring, UK) and group 2 will receive oxytocin 5IU (Syntocinon®, Novartis, Switzerland).

DETAILED DESCRIPTION:
Obstetric haemorrhage remains one of the major causes of maternal death in both developed and developing countries. Postpartum haemorrhage (PPH) is defined as a blood loss >500 ml more of blood from the genital tract within 24 hours of the birth of a baby. PPH can be minor (500-1000 ml) or major (more than 1000 ml) . The most frequent cause of PPH is uterine atony, contributing up to 80 % of the PPH cases.

Risk factors of atonic PPH include multiple pregnancy, placenta previa, previous PPH, body mass index (BMI) >30, prolonged labour, fetal macrosomia>4kg and primipara> 40 years.

Placenta praevia exists when the placenta is inserted wholly or in part into the lower segment of the uterus. It is classified by ultrasound imaging according to what is relevant clinically: if the placenta lies over the internal cervical os, it is considered a major praevia; if the leading edge of the placenta is in the lower uterine segment but not covering the cervical os, minor or partial praevia exists.

Oxytocin is currently the uterotonic of first choice. It has proven to decrease the incidence of PPH by 40 % and has a rapid onset of action and a good safety profile. A disadvantage of oxytocin is its short half-life of 4-10 min, regularly requiring a continuous intravenous infusion or repeated intramuscular injections.

Carbetocin is a long-acting oxytocin analogue indicated for the prevention of uterine atony after child birth by cesarean section (CS) under epidural or spinal anaesthesia. Carbetocin has a rapid onset of action (within 1-2 min) and a prolonged duration of action (approximately 1 h) because of sustained uterine response with contractions of higher amplitude and frequency. Its safety profile is comparable to that of oxytocin.

The study will be conducted in Cairo university hospitals and BeniSuef university hospitals. All patients with placenta previa covering, or less than 2cm from the internal cervical os will be approached in the antenatal clinic. Women will be invited to participate in the study, the invitation will include a clear full explanation of the study. Only patients signing informed written consents will participate in the study.

The exclusion criteria will be gestational age <37 weeks, hypertension, preeclampsia, cardiac, renal or liver diseases, epilepsy, need for general anaesthesia, known hypersensitivity to carbetocin and suspected placenta accreta.

200 women will be randomly divided into 2 equal groups using computer generated random numbers, Group 1 will receive Carbetocin 100 µgm (Pabal® Ferring, UK) and group 2 will receive oxytocin 5IU (Syntocinon®, Novartis, Switzerland). Both drugs will be diluted in 10ml saline and will be given by the anaesthetist slowly intravenously after delivery of the baby. The investigators will not include a control group for ethical reasons.

The CS will be done in the presence of a consultant Obstetrician and a consultant anaesthetist, cross-matched blood will be ready and a level 2 critical care bed will be available. CS will be done through the lower uterine segment, if the placenta is encountered, it will be pushed aside and the baby will be delivered.

The allocated drug will be diluted in 10ml saline and will be given by the anesthesist slowly intravenously after delivery of the baby. The uterine tone and amount of bleeding will be noted and the need for further uterotonic agents will be determined 2 minutes after giving the drug.

Blood loss will be estimated through weighing the swabs, using pictorial charts and estimating the amount of blood in the suction containers. Blood haemoglobin will be assessed 24 hours after the CS.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing CS for placenta previa

Exclusion Criteria:

* Gestational age <37 weeks
* Hypertension
* Preeclampsia
* Cardiac, renal or liver diseases
* Need for general anaesthesia
* Known hypersensitivity to carbetocin
* Suspected placenta accreta

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Need for other uterotonic drugs | 2 minutes after giving the drug
  If the uterus is not contracted 2 minutes after giving the drug, further uterotonic drugs will be given.

SECONDARY OUTCOMES:
Development of PPH | 2 minutes after giving the drug.
  PPH will be diagnosed when bleeding exceeds 500ml

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - BeniSuef University hospitals, BeniSuef
  - Cairo university hospitals, Cairo

REFERENCES:
- [Background] Moertl MG, Friedrich S, Kraschl J, Wadsack C, Lang U, Schlembach D. Haemodynamic effects of carbetocin and oxytocin given as intravenous bolus on women undergoing caesarean delivery: a randomised trial. BJOG. 2011 Oct;118(11):1349-56. doi: 10.1111/j.1471-0528.2011.03022.x. Epub 2011 Jun 14. PMID 21668768
- [Result] Winter C, Macfarlane A, Deneux-Tharaux C, Zhang WH, Alexander S, Brocklehurst P, Bouvier-Colle MH, Prendiville W, Cararach V, van Roosmalen J, Berbik I, Klein M, Ayres-de-Campos D, Erkkola R, Chiechi LM, Langhoff-Roos J, Stray-Pedersen B, Troeger C. Variations in policies for management of the third stage of labour and the immediate management of postpartum haemorrhage in Europe. BJOG. 2007 Jul;114(7):845-54. doi: 10.1111/j.1471-0528.2007.01377.x. PMID 17567419